CLINICAL TRIAL: NCT00878709
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Of Neratinib (HKI-272) After Trastuzumab In Women With Early-Stage HER-2/Neu Overexpressed/Amplified Breast Cancer
Brief Title: Study Evaluating The Effects Of Neratinib After Adjuvant Trastuzumab In Women With Early Stage Breast Cancer
Acronym: ExteNET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3144A2-3004 / B1891004
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: HER-2/erbB-2 positive breast cancer; breast cancer; adjuvant therapy; neratinib; HKI-272; Nerlynx; PB-272
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neratinib (Experimental): 240 mg orally daily for one year
  Interventions: Drug: neratinib
- Placebo (Placebo Comparator): orally daily for one year
  Interventions: Other: placebo

INTERVENTIONS:
Drug: neratinib
  Other Names: HKI-272; Nerlynx
  Arms: Neratinib
Other: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether neratinib can further reduce the risk of recurrence from previously diagnosed HER-2 positive breast cancer after adjuvant treatment with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Stage II through IIIC HER-2/erbB-2 positive breast cancer with node positive disease.
* Been treated for early breast cancer with standard of care duration of trastuzumab.
* Could have been treated neoadjuvantly but have not reached pathologic complete response.

Exclusion Criteria:

* Positive clinical and radiologic assessments for local or regional recurrence of disease at the time of study entry.
* History of heart disease.
* Corrected QT (QTc) interval >0.45 seconds
* History of gastrointestinal disease with diarrhea as the major symptom.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2840 (Actual)
Dates: Start 2009-07-09 (Actual); Primary Completion 2014-08-21 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Vice President Clinical Science and Pharmacology, Study Director — Puma Biotechnology, Inc.
Locations (493):
- United States (185):
  - Anniston Oncology, Anniston, Alabama
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - NAHOA, Sedona, Arizona
  - Arizona Oncology Associates, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Cedars-Sinai Medical Group, Beverly Hills, California
  - Ronald Yanagihara, M.D., Gilroy, California
  - Glendale Adventist Medical Center Cancer Services, Glendale, California
  - California Cancer Care, Greenbrae, California
  - Beaver Medical Group, L.P., Highland, California
  - Breastlink Medical Group, Long Beach, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Facey Medical Group, Mission Hills, California
  - Gynecologic Oncology Associates, Newport Beach, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Desert Hematology Oncology Medical Group, Inc, Rancho Mirage, California
  - Helen Diller Family University of California San Francisco Comprehensive Cancer Center, San Francisco, California
  - San Francisco Oncology Associates, San Francisco, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - The Cancer Prevention and Treatment Center, Soquel, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Hematology Oncology, PC, Stamford, Connecticut
  - Connecticut Oncology and Hematology, Torrington, Connecticut
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Innovative Medical Research of South Florida, Inc., Aventura, Florida
  - University Cancer Institute, LLC, Boynton Beach, Florida
  - North Broward Medical Center, Deerfield Beach, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Florida Cancer Specialists and Research Institute, Gainesville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Hematology Oncology Associates, Loxahatchee Groves, Florida
  - Florida Cancer Affiliates - Ocala, Ocala, Florida
  - Mid-Florida Hematology & Oncology Centers, PA, Orange City, Florida
  - Cancer Centers of Florida, Orlando, Florida
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Florida Cancer Research Institute, Plantation, Florida
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists, P.L., St. Petersburg, Florida
  - Oncology and Hematology of West Broward, Tamarac, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Phoebe Cancer Center, Albany, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Augusta Oncology Associates (ACORN), P.C., Augusta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Straub Clinic & Hospital, Honolulu, Hawaii
  - Portneuf Medical Center, Pocatello, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois, Decatur Memorial Hospital Clinical Research, Decatur, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Medical Arts Associates, Ltd, Moline, Illinois
  - Advocate Medical Group, Niles, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, Niles, Illinois
  - Quincy Medical Group, Cancer Center at Blessing Hospital, Quincy, Illinois
  - North Shore Cancer Research Associates, Skokie, Illinois
  - Orchard Healthcare Research, Inc., Skokie, Illinois
  - Orchard Research, LLC, Skokie, Illinois
  - Simmons Cancer Institute, Springfield, Illinois
  - Springfield Clinic, LLP, Springfield, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Hematology Oncology of Indiana, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - Purchase Cancer Group, Paducah, Kentucky
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - Crescent City Research Consortium, LLC, Marrero, Louisiana
  - Central Maine Healthcare Corp, Lewiston, Maine
  - Mercy Hospital Oncology/Hematology Center, Portland, Maine
  - York Hospital Oncology Treatment Center, York Village, Maine
  - Medical Oncology & Hematology Mercy Medical Center, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Center, Baltimore, Maryland
  - Alliance Hematology Oncology, PA Carroll County Cancer Center, Westminster, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital - Gillette Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Medical Specialty Associates, Grand Rapids, Michigan
  - Northern Michigan Hematology/Oncology, Petoskey, Michigan
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - North Mississippi Hematology and Oncology Associates, Ltd., Tupelo, Mississippi
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - St. Joseph's Oncology, Saint Joseph, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Montana Cancer Specialists, Missoula, Montana
  - Southeast Nebraska Hematology & Oncology Consultants, PC, Lincoln, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Trinitas Comprehensive Cancer Center, Elizabeth, New Jersey
  - Saint Barnabas Health Care System, Livingston, New Jersey
  - Summit Medical Group, Morristown, New Jersey
  - Oncology and Hematology Specialist, Mountain Lakes, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - The Valley Hospital, Luckow Pavilion, Paramus, New Jersey
  - Cooper University Hospital, Voorhees Township, New Jersey
  - ProHealth Care Associates, Lake Success, New York
  - NYU Clinical Cancer Center, New York, New York
  - Columbia University Medical Center, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - NorthEast Oncology Associates Carolinas Medical Center NorthEast, Concord, North Carolina
  - Duke University Medical Center Medical Oncology, Durham, North Carolina
  - Raleigh Hematology Oncology Associates Cancer Centers of North Carolina, Raleigh, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Signal Point Hematology/Oncology, Inc., Middletown, Ohio
  - Mercy Physicians of Oklahoma, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Samaritan Hematology & Oncology Consultants, Corvallis, Oregon
  - Northwest Cancer Specialist, P.C., Portland, Oregon
  - Providence Cancer Center Oncology and Hematology Care - Westside, Portland, Oregon
  - Kaiser Permanente Northwest Region Oncology Hematology, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Oncology-Hematology of Lehigh Valley, PC, Bethlehem, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Pinnacle Health Cancer Center Community Campus, Harrisburg, Pennsylvania
  - Sweeney-Melenyser Pavillion, Monongahela, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Clinic, Limited, Sayre, Pennsylvania
  - Abington Hematology Oncology Associates, Inc, Willow Grove, Pennsylvania
  - Pawtuket Memorial Hospital, Pawtucket, Rhode Island
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - Francisco Gonzalez MD PA, Columbia, South Carolina
  - McLeod Oncology and Hematology Associates, Florence, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - Santee Hematology Oncology, Sumter, South Carolina
  - Avera Medical Oncology and Hematology - Avera Cancer Institute, Sioux Falls, South Dakota
  - University Hematology/Oncology Associates PLLC, Chattanooga, Tennessee
  - Cookeville Regional Cancer Center, Cookeville, Tennessee
  - The Jones Clinic, PC, Germantown, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - South Texas Institute of Cancer, Corpus Christi, Texas
  - Cancer Specialists of South Texas, P.A., Corpus Christi, Texas
  - Center for Oncology Research, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center Simmons Cancer Center, Dallas, Texas
  - Texas Oncology, P.A., Denton, Texas
  - El Paso Cancer Treatment Center - West, El Paso, Texas
  - Center for Integrative Cancer Medicine, PA, El Paso, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, P.A., Garland, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - The Methodist Hospital Breast Center, Houston, Texas
  - Medicus Alliance Clinical Research Org., Inc., Houston, Texas
  - Jabboury Foundation for Cancer Research, Inc., Houston, Texas
  - Texas Oncology, P.A., Paris, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - South Texas Oncology & Hematology, San Antonio, Texas
  - Texas Oncology P.A., Sugar Land, Texas
  - East Texas Medical Center Cancer Institute, Tyler, Texas
  - Texas Oncology, Tyler, Texas
  - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - North Utah Associates, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Rutland Regional Medical Center, Rutland, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Cascade Cancer Center, Kirkland, Washington
  - Cancer Care Northwest-North, Spokane, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - West Virginia University Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Wheaton Franciscan Cancer Care-All Saints, Racine, Wisconsin
- Australia (8):
  - Sydney West Cancer Trials Centre, Sydney, New South Wales
  - Iron Cancer Care South Brisbane, South Brisbane, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - North Adelaide Oncology Calvary Hospital North Adelaide, North Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
  - The Western Hospital, Melbourne, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
- Belgium (13):
  - OLVZ Medische Oncologie, Aalst
  - Az. St. Jan, Bruges
  - Cliniques Universitaires de Bruxelles, Brussels
  - VZW Jesseziekenhuis - Campus Virga Jesse, Hasselt
  - Jan Yperman Ziekenhuis, Ieper
  - AZ Groeninge ampus Maria's Voorzienigheid (MV) Oncologisch Centrum, Kortrijk
  - Centre Hospitalier Regional de La Citadelle, Liège
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
  - C.H.U. Ambroise Paré, Mons
  - AZ Damiaan - Site Sint-Jozef, Ostend
  - AZ Zusters van Barmhartigheid, Ronse
  - AZ Nikolaas, Sint-Niklaas
  - Sint-Elisabethziekenhuis, Turnhout
- Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil
- Bulgaria (5):
  - District Dispensary for Oncology Diseases Internal Unit- Plovdiv EOOD, Ist, Plovdiv
  - District Dispensary for Oncology Diseases Internal Unit- Plovdiv EOOD, Second, Plovdiv
  - District Dispensary for Oncology Diseases Internal Unit- Sofia EOOD, Sofia
  - Specialised Hospital of Active Treatment in Oncology, Sofia
  - Interdistrict Dispensary for Oncology Diseases, Varna
- Canada (14):
  - Cross Cancer Institute, Edmonton, Alberta
  - Jack Ady Cancer Centre, Lethbridge, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Cancer Centre at Southlake, Newmarket, Ontario
  - R.S. McLaughlin Durham Regional Cancer Centre, Oshawa, Ontario
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital - Church Street Site, Weston, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - C.H.U.M. - Hopital Notre-Dame, Departement d'Oncologie, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire de Quebec Hopital du St-Sacrement, Québec, Quebec
  - CSSS Alphonse-Desjardins, Québec, Quebec
- China (9):
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital of Chinese Academy of Medical Sciences, Beijing
  - The Hospital Affiliated Academy Military Medical Science, Chinese People's, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Southern Medical University Nanfang Hospital, Guangzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
- Colombia (3):
  - Oncomedica S.A. IMAT, Montería, Departamento de Córdoba
  - Oncologos del Occidente, Pereira, Risaralda Department
  - Administradora Country S.A-Clinica del Country, Bogotá
- Croatia (4):
  - University Hospital Centre Osijek, Department of Radiotherapy and Oncology, Osijek
  - General Hospital Varazdin, Varaždin
  - Klinicki bolnicki centar "Sestre Milosrdnice", Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (6):
  - Fakultni nemocnice Brno, Brno
  - Masarykuv Onkologicky ustav, Brno
  - Nemocnice Jihlava, Jihlava
  - Institut Onkologie a Reahabilitace na Plesi, Nová Ves pod Pleší
  - Multiscan s. r. o., Pardubice
  - Fakultni Nemocnice v Motole, Prague
- Denmark (12):
  - Aalborg Sygehus, Aalborg
  - Aarhus University Hospital, Aarhus C
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg
  - Herlev Hospital, Herlev
  - Hillerod Hospital, Hillerød
  - Næstved Sygehus, Næstved
  - Odense Universitetshospital, Odense C
  - Roskilde University Hospital, Roskilde
  - Sygehus Sonderjylland, Sønderborg
  - Vejle Sygehus, Vejle
  - Regionshospital Viborg, Viborg
- France (20):
  - Centre Rene Gauducheau, Saint-Herblain, Cedex
  - C.H.U. De Bordeaux Saint Andre, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Hospitalier de Montluçon, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Oncologie department, Hopital albert Michalon, Grenoble
  - Hopital de Versailles, Le Chesnay
  - Centre Oscar Lambret, Lille
  - Institut Curie, Département d'Oncologie Médicale, Paris
  - Hopital Saint Louis, Paris
  - Hopital La Pitie-Salpetriere, Paris
  - Service d'Oncologie et de Radiotherapie, Polyclinique Francheville, 38, Périgueux
  - Centre Henri Becquerel, Rouen
  - Pole Hospitalier Mutualiste, Saint-Nazaire
  - Institute de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Clinique Sainte Anne Centre de Radiothérapie, Strasbourg
  - CHU Strasbourg, Strasbourg
  - CHU Bretonneau Centre Henry Kaplan, Tours
  - Institut Gustave Roussy, Villejuif
  - CHU Paul Brousse, Villejuif
- Germany (36):
  - Marienhospital, Aachen
  - Onkologische Praxis, Augsburg
  - Sozialstiftung Bamberg Klinik fuer Haematologie und Internistische Onkologie, Bamberg
  - Onkologische Schwerpunktpraxis, Berlin
  - Praxisklinik Krebsheilkunde fuer Frauen, Berlin
  - Frauenarzt-Zentrum-Zehlendorf, Berlin
  - Universitaetsklinikum Duesseldorf, Frauenklinik, Düsseldorf
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Luisenkrankenhaus, Düsseldorf
  - Facharzt fuer Frauenheilkunde und Geburtshilfe, Erfurt
  - Onkologische Gemeinschaftspraxis Frankfurt, Frankfurt am Main
  - Frauenklinik der J.W. Goethe-Universitaet, Frankfurt am Main
  - Staedtische Kliniken Frankfurt am Main-Hoechst Frauenklinik, Frankfurt am Main
  - Praxis für interdisziplinaere Onkologie & Haematologie GbR, Freiburg im Breisgau
  - Klinikum St. Georg/Franziskus, Abteilung fuer Senologie, Georgsmarienhütte
  - Kreiskrankenhaus Hameln, Onkologische Ambulanz, Hamelin
  - Facharzt fuer Frauenheilkunde, Hanover
  - Onkologische Schwerpunktpraxis, Heidelberg
  - Nationales Centrum fuer Tumorerkrankungen, Heidelberg
  - Klinikum Kempten - Oberallgaeu, Kempten
  - MTV Abts & Partner Kiel, Kiel
  - Universitaetsfrauenklinikum Schleswig-Holstein, Lübeck
  - Universitaetsklinikum Magdeburg A.oe.R., Magdeburg
  - Klinikum der Johannes-Gutenberg-Universitaet, Mainz
  - Fachpraxis fuer Innere Medizin, München
  - Klinik und Poliklinik fuer, München
  - Praxis Gynaekologie Arabella Muenchen, München
  - Klinik fuer Gynaekologie und Geburtshilfe, Offenbach
  - Pius-Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg GmbH, Oldenburg
  - Oncologianova GmbH, Recklinghausen
  - Universitaetsfrauenklinik Tuebingen, Tübingen
  - St. Marienhospital Vechta, Vechta
  - Gemeinschaftspraxis fuer Haematologie und Onkologie, Westerstede
  - Klinik für Gynaekologie und gyn. Onkologie, Wiesbaden
  - Marienhospital Witten, Witten
- Greece (8):
  - University Hospital of Heraklion, Heraklion, Creete
  - General Hospital of Chania Ag. Georgios, Chania, Crete
  - University General Hospital of Alexandroupoli, Department of Medical Oncology, Alexandroupoli
  - Hippokratio General Hospital of Athens, Athens
  - Hippokration Hospital Athens, Athens
  - University General Hospital of Larissa, Larissa
  - University Hospital of Patras, Rio Patras
  - Euromedica General Clinic, Thessaloniki
- Hong Kong (5):
  - UNIMED Medical Institute, Comprehensive Centre for Breast Diseases, Hong Kong, Wan Chai
  - Department of Clinical Oncology, Tuen Mun Hospital, Hong Kong
  - Queen Mary Hospital, Department of Clinical Oncology, Professorial Block, Hong Kong
  - Queen Mary Hospital, Department of Medicine, Blk K, Hong Kong
  - Queen Mary Hospital, Department of Medicine, Hong Kong
- Hungary (9):
  - Semmelweis Egyetem Radiologiai és Onkoterapias Klinika, Budapest
  - Fovarosi Onkormanyzat Szent Imre Korhaz, Budapest
  - Orszagos Onkologiai Intezet "B" Belgyogyaszati osztaly, Budapest
  - Bekes M. Kepviselotest. Pandy Kalman Korhaz, Megyei Onkol. Kp., Klin. Onkol. es Sugartherapias Oszt., Gyula
  - Kaposi Mor Oktato Korhaz, Onkologiai Centrum, Kaposvár
  - Bacs-Kiskun Megyei Korhaz Onkoradiologiai Kozpont, Kecskemét
  - Borsod-Abauj-Zemplen M. Korhaz es Egyetemi Okt. K., Klin. Onk., Sugarterapias es Kozp. Szuro Centrum, Miskolc
  - Josa Andras Oktatokorhaz Egeszsegugyi Szolgaltato Nonprofit Kft. / Onkoradiologiai Osztaly, Nyíregyháza
  - Veszprem Megyei Csolnoky Ferenc Korhaz Nonprofit Zrt., Veszprém
- Israel (4):
  - Soroka University MC, Department of Oncology, Beersheba
  - Rambam Health care campus, Oncology institute, Haifa
  - Kaplan Medical Center, Department of Oncology, Rehovot
  - Sheba Medical Center, Oncology Institute Tel Hashomer, Tel Litwinsky
- Italy (19):
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Presidio Ospedaliero di Summa - Antonio Perrino, Brindisi
  - Azienda Ospedaliera Universitaria "Policlinico Vittorio Emanuele", Catania
  - Fondazione per la Ricerca e la Cura dei Tumori Tommaso Campanella, Catanzaro
  - Azienda Ospedaliera San Gerardo, Monza
  - Fondazione Giovanni Pascale, Napoli
  - Unita' Operativa Complessa Oncologia Medica, A.O.R.N. "Cardarelli", Napoli
  - Azienda Ospedaliera San Luigi Gonzaga, Orbassano (TO)
  - IRCCS Istituto Oncologico Veneto di Padova, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Universita Campus Bio-Medico, Roma
  - Oncologia Medica A, Istituti Fisioterapici Ospitalieri, Roma
  - Ospedale San Pietro Fatebenefratelli, Roma
  - Ospedale SS Trinita, Sora (FR)
  - Azienda Ospedaliera S. Maria, Terni
  - Ospedale Treviglio e Caravaggio, UO Oncologia Medica, Treviglio, BG
  - Istituto Oncologico del Mediterraneo, Viagrande (CT)
  - Ospedale Belcolle Viterbo, Viterbo
- Japan (23):
  - Aichi Cancer Center, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kurume Daiichi Social Insurance Hospital, Fukuoka
  - Hiroshima City Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hyogo Cancer Center, Hyōgo
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kumamoto Municipal Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Niigata Cancer Center Hospital 2-15-3, Niigata
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - Tokyo Metropolitan Cancer and Infectious disease Center Komagome Hp, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo
- Lithuania (2):
  - The Hospital of Lithuanian University of Health Sciences Kauno klinikos Oncology and Haematology Clinic, Kaunas
  - Oncology Institute of Vilnius University, Vilnius
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Sir Paul Boffa Hospital, Floriana, Malta
- Nucleo de Especialidades Oncológicas, Guadalajara, Jalisco, Mexico
- Netherlands (7):
  - Ziekenhuis Amstelland, Amstelveen
  - Gelre ZH, Apeldoorn
  - Amphia Ziekenhuis - Interne Geneeskunde, Breda
  - Maxima Medisch Centrum, Eindhoven
  - Vlietland Ziekenhuis, Schiedam
  - Orbis Medisch Centrum, Sittard-Geleen
  - Haga Ziekenhuis, The Hague
- Auckland Hospital, Auckland, New Zealand
- University Clinic for Radiotherapy and Oncology, Skopje, North Macedonia
- Clínica Vista Alegre / Unidad de Investigacion, Surco, Lima region, Peru
- Poland (11):
  - Bialostockie Centrum Onkologii im. M. Sklodowskiej- Curie w Bialymstoku, Bialystok
  - Centrum Onkologii im. prof. Franciszka Łukaszczyka, Bydgoszcz
  - Centrum Medyczne Ostrobramska Niepubliczny Zaklad Opieki Zdrowotnej "Magodent", Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne w Gdansku, Gdansk
  - Szpital Morski im. PCK Gdynskie Centrum Onkologii Oddzial Chemioterapii, Gdynia
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Wojewodzki Oddzial, Jelenia Góra
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w, Krakow
  - Zaklad Opieki Zdrowotnej MSWiA z Warminsko - Mazurskim Centrum Onkologii w, Olsztyn
  - Olsztynski Osrodek Onkologiczny Kopernik Sp. z o.o., Olsztyn
  - Szpital Wojewodzki im. Sw. Lukasza Samodzielny Publiczny Zaklad Opieki, Tarnów
  - Centrum Medyczne Ostrobramska Niepubliczny Zaklad Opieki Zdrowotnej "Magodent", Warsaw
- Romania (3):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta", Cluj-Napoca, Cluj
  - SC Oncolab S.R.L., Craiova, Dolj
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
- Serbia (2):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Clinical centre Nis, Niš
- National Cancer Centre Singapore, Singapore, Singapore
- Slovakia (3):
  - Interna onkologicka klinika, Bratislava
  - Oddelenie radioterapie a onkologie, Košice
  - Poliklinika ADUS, Poprad
- South Korea (5):
  - Samsung Medical Center, Seoul, Korea
  - National Cancer Center, Center for Breast Cancer, Gyeonggi-do
  - Seoul National University Hospital, Department of Internal Medicine, Seoul
  - Korea University Anam Hospital, Department of Oncology/Hematology, Seoul
  - Asan Medical Center, Seoul
- Spain (36):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de Torrevieja, Torrevieja, Alicante
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO de Barcelona - Hospital Duran i Reynals, Hospitalet de Llobregat Consorci Sanitari de Terrassa, L'Hospitalet de Llobregat, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
  - Hospital de Barbastro, Barbastro, Huesca
  - Hospital Universitario Fundacion de Alcorcon, Alcorcón, Madrid
  - Hospital Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital De Basurto, Bilbao, Vizcaya
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Universitario Vall D´Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - ICO de Girona - Hospital Universitario de Girona Dr. Josep Trueta, Girona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Madrid Norte Sanchinarro. Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Clinico Universitario Virgen de La Victoria, Málaga
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Virgen de la Salud, Toledo
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Provincial de Zamora, Zamora
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Onkologiska Kliniken, Lund
  - Skanes Onkologiska Kliniken, Lund
- Switzerland (4):
  - Hirslanden Medical Center Tumor Center, Aarau
  - Kantonsspital Baden, Baden
  - Kantonsspital Olten-Medizinische Onkologie, Olten
  - Spital STS AG, Thun
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Linkou Branch, Kwei-Shan, Taoyuan
  - National Taiwan University Hospital, Taipei TOC
- Affinity Research Limited, Nassau, The Bahamas
- Turkey (Türkiye) (10):
  - Gazi Universitesi Tip Fakultesi, Besevler/Ankara
  - Ege Universitesi Tip Fakultesi, Bornova/Izmir
  - Istanbul Universitesi Istanbul Tip Fakultesi, Capa/Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Ic Hastaliklari Anabilim Dali, Cerrahpasa/Istanbul
  - Dr. Abdurrahman Yurtaslan Onkoloji Egitim ve Arastirma Hastanesi, Demetevler/Ankara
  - Uludag Universitesi Tip Fakultesi, Gorukle/Bursa
  - Dokuz Eylul Universitesi Tip Fakultesi, Inciralti/Izmir
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Gaziantep Universitesi, Sehitkamil/Gaziantep
  - Hacettepe Universitesi Tip Fakultesi, Sihhiye/Ankara
- United Kingdom (13):
  - Betsi Cadwaladr University Health Board, Rhyl, Denbighshire
  - Queens Hospital, Burton-on-Trent, Staffs
  - St James's University Hospital, Leeds
  - University Hospitals of Leicester, Leicester
  - St. Bartholomew's Hospital, London
  - Guy's Hospital, London
  - Charing Cross Hospital, Department Of Medical Oncology, London
  - Christie Hospital, Manchester
  - Norfolk & Norwich University Hospitals, Norwich
  - Nottingham City Hospital, Nottingham
  - Weston Park Hospital, Sheffield
  - Singleton Hospital, Swansea
  - Southend University Hospital, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Puma Biotechnology is committed to sharing clinical trial data and information to help physicians and patients make informed treatment decisions, and to help qualified researchers advance scientific knowledge.
  In accordance with legal and regulatory requirements, Puma publishes study protocol information and clinical study results on clinical trial registries, including ClinicalTrials.gov and EU Clinical Trials Register. Puma also publishes information about clinical studies in peer-reviewed scientific journals and shares data in scientific meetings.
  Puma commits to safeguarding confidentiality and patient privacy throughout the clinical trial data and information sharing process. Any patient-level data will be anonymized to protect personally identifiable information.
  Qualified researchers and study participants may submit requests for other study documentation and clinical trial data to clinicaltrials@pumabiotechnology.com for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Clinical study documents and clinical trial data may be requested by qualified researchers and study participants for studies that have been completed for at least 18 months, and for which the indication of the drug has been approved in the US and/or EU, as applicable. Requests will be accepted for up to 24 months after the criteria described in this section are met.
Access Criteria: Requestors must provide organizational contact information; a detailed research plan, including outcomes; timeline for completion of the research; qualifications of the research team; funding source; and potential conflicts of interest.
  Puma will not provide access to patient-level data if there is a reasonable likelihood that individual patients could be identified, or in cases where confidentiality or consent provisions prohibit transfer of data or information to third parties. Additionally, Puma will not disclose information that jeopardizes intellectual property rights or divulges confidential commercial information.
URL: https://pumabiotechnology.com/data_sharing_policy.html

REFERENCES:
- [Derived] Holmes FA, Moy B, Delaloge S, Chia SKL, Ejlertsen B, Mansi J, Iwata H, Gnant M, Buyse M, Barrios CH, Silovski T, Separovic R, Bashford A, Zotano AG, Denduluri N, Patt D, Gokmen E, Gore I, Smith JW 2nd, Loibl S, Masuda N, Tomasevic Z, Petrakova K, DiPrimeo D, Wong A, Martin M, Chan A; ExteNET Study Group. Overall survival with neratinib after trastuzumab-based adjuvant therapy in HER2-positive breast cancer (ExteNET): A randomised, double-blind, placebo-controlled, phase 3 trial. Eur J Cancer. 2023 May;184:48-59. doi: 10.1016/j.ejca.2023.02.002. Epub 2023 Feb 10. PMID 36898233
- [Derived] Iwata H, Masuda N, Kim SB, Inoue K, Rai Y, Fujita T, Chiu J, Ohtani S, Takahashi M, Miyaki T, Lu YS, Xu B, Yap YS, Bustam A, Yao B, Zhang B, Bryce R, Chan A. Neratinib after trastuzumab-based adjuvant therapy in patients from Asia with early stage HER2-positive breast cancer. Future Oncol. 2019 Jul;15(21):2489-2501. doi: 10.2217/fon-2019-0143. Epub 2019 May 29. PMID 31140297
- [Derived] Chia SKL, Martin M, Holmes FA, Ejlertsen B, Delaloge S, Moy B, Iwata H, von Minckwitz G, Mansi J, Barrios CH, Gnant M, Tomasevic Z, Denduluri N, Separovic R, Kim SB, Jakobsen EH, Harvey V, Robert N, Smith J 2nd, Harker G, Zhang B, Eli LD, Ye Y, Lalani AS, Buyse M, Chan A. PIK3CA alterations and benefit with neratinib: analysis from the randomized, double-blind, placebo-controlled, phase III ExteNET trial. Breast Cancer Res. 2019 Mar 11;21(1):39. doi: 10.1186/s13058-019-1115-2. PMID 30867034
- [Derived] Mortimer J, Di Palma J, Schmid K, Ye Y, Jahanzeb M. Patterns of occurrence and implications of neratinib-associated diarrhea in patients with HER2-positive breast cancer: analyses from the randomized phase III ExteNET trial. Breast Cancer Res. 2019 Feb 27;21(1):32. doi: 10.1186/s13058-019-1112-5. PMID 30813966
- [Derived] Delaloge S, Cella D, Ye Y, Buyse M, Chan A, Barrios CH, Holmes FA, Mansi J, Iwata H, Ejlertsen B, Moy B, Chia SKL, Gnant M, Smichkoska S, Ciceniene A, Martinez N, Filipovic S, Ben-Baruch NE, Joy AA, Langkjer ST, Senecal F, de Boer RH, Moran S, Yao B, Bryce R, Auerbach A, Fallowfield L, Martin M. Effects of neratinib on health-related quality of life in women with HER2-positive early-stage breast cancer: longitudinal analyses from the randomized phase III ExteNET trial. Ann Oncol. 2019 Apr 1;30(4):567-574. doi: 10.1093/annonc/mdz016. PMID 30689703
- [Derived] Martin M, Holmes FA, Ejlertsen B, Delaloge S, Moy B, Iwata H, von Minckwitz G, Chia SKL, Mansi J, Barrios CH, Gnant M, Tomasevic Z, Denduluri N, Separovic R, Gokmen E, Bashford A, Ruiz Borrego M, Kim SB, Jakobsen EH, Ciceniene A, Inoue K, Overkamp F, Heijns JB, Armstrong AC, Link JS, Joy AA, Bryce R, Wong A, Moran S, Yao B, Xu F, Auerbach A, Buyse M, Chan A; ExteNET Study Group. Neratinib after trastuzumab-based adjuvant therapy in HER2-positive breast cancer (ExteNET): 5-year analysis of a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1688-1700. doi: 10.1016/S1470-2045(17)30717-9. Epub 2017 Nov 13. PMID 29146401
- [Derived] Chan A, Delaloge S, Holmes FA, Moy B, Iwata H, Harvey VJ, Robert NJ, Silovski T, Gokmen E, von Minckwitz G, Ejlertsen B, Chia SKL, Mansi J, Barrios CH, Gnant M, Buyse M, Gore I, Smith J 2nd, Harker G, Masuda N, Petrakova K, Zotano AG, Iannotti N, Rodriguez G, Tassone P, Wong A, Bryce R, Ye Y, Yao B, Martin M; ExteNET Study Group. Neratinib after trastuzumab-based adjuvant therapy in patients with HER2-positive breast cancer (ExteNET): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):367-377. doi: 10.1016/S1470-2045(15)00551-3. Epub 2016 Feb 10. PMID 26874901

RESULTS

PARTICIPANT FLOW:
Groups:
- Neratinib: Patients who completed prior adjuvant trastuzumab received six 40 mg neratinib tablets (240 mg) taken orally once daily with food, preferably in the morning, continuously for one year. Therapy continued until unacceptable toxicity, recurrent disease, death, or withdrawal of consent occurred.
- Placebo: Patients who completed prior adjuvant trastuzumab received six 40 mg placebo tablets (240 mg) taken orally once daily with food, preferably in the morning, continuously for one year.Therapy continued until unacceptable toxicity, recurrent disease, death, or withdrawal of consent occurred.
Period: Overall Study
Arm/Group | Neratinib | Placebo
Started | 1420 | 1420
Completed | 1095 | 1183
Not Completed | 325 | 237
Not completed — Withdrawal by Subject | 197 | 120
Not completed — Lost to Follow-up | 35 | 33
Not completed — Other Reasons | 93 | 84

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants who were randomized regardless of whether they received any study treatment.
Groups:
- Placebo: Patients who completed prior adjuvant trastuzumab received six 40 mg placebo tablets (240 mg) taken orally once daily with food, preferably in the morning, continuously for one year. Therapy continued until unacceptable toxicity, recurrent disease, death, or withdrawal of consent occurred.
- Total: Total of all reporting groups
Arm/Group | Neratinib | Placebo | Total
Number analyzed (Participants) | 1420 | 1420 | 2840
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.08) | 52.3 (10.28) | 52.3 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1420 | 1420 | 2840
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 188 | 197 | 385
  Black or African American | 27 | 47 | 74
  White | 1165 | 1135 | 2300
  Other | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-free Survival (iDFS) in Neratinib Arm Compared to Placebo Arm at Year 2
Description: Invasive disease-free survival time is defined as the time from date of randomization until the first disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, distant recurrence and death from any cause.
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 4.7 | 7.5
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Invasive disease-free survival (iDFS) in neratinib arm compared to placebo arm; Test type: Superiority; p = 0.008, Log Rank; The Log-rank test is stratified by prior trastuzumab (concurrent or sequential), nodal status (<= 3 or >= 4) and ER/PgR status (positive or negative); Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.49 to 0.90] — The hazard ratio is estimated by stratified Cox model. The Cox model is stratified by prior trastuzumab (concurrent or sequential), nodal status (<= 3 or >= 4) and ER/PgR status (positive or negative)

2. Primary Outcome: Kaplan-Meier Estimates of Invasive Disease-free Survival (iDFS) at Year 2 by Treatment Arms
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants | 94.2 [92.6 to 95.4] | 91.9 [90.2 to 93.2]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause, censored at the last date known alive.
Time Frame: Randomization until death due to any cause (up to 119 Months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants
  1 Year Kaplan-Meier Estimate | 99.64 [99.13 to 99.85] | 99.43 [98.86 to 99.71]
  3 Year Kaplan-Meier Estimate | 96.74 [95.62 to 97.57] | 96.44 [95.30 to 97.31]
  5 Year Kaplan-Meier Estimate | 94.09 [92.65 to 95.25] | 93.26 [91.77 to 94.49]
  7 Year Kaplan-Meier Estimate | 91.36 [89.66 to 92.79] | 91.29 [89.62 to 92.70]
  9 Year Kaplan-Meier Estimate | 89.06 [86.97 to 90.84] | 88.65 [88.58 to 90.43]
Statistical Analysis 1: Comparison: Neratinib vs Placebo; The 2-sided P-value was based on stratified log-rank test (stratification factors: prior Trastuzumab (concurrent or sequential), nodal status (<=3 or >=4) and ER/PgR status (positive or negative). The hazard ratio and corresponding 95% CI from the stratified cox proportional hazard model were also presented; Test type: Superiority; p = 0.6914, Log Rank; Hazard Ratio (HR) = 0.952, 95% CI 2-sided [0.747 to 1.212]

4. Secondary Outcome: Disease-free Survival Including Ductal Carcinoma in Situ (DFS-DCIS) in Neratinib Arm Compared to Placebo Arm at Year 2
Description: Disease-free survival including DCIS time is defined as the time from date of randomization until the first occurrence of DCIS or an iDFS event (an iDFS event including invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, or distant recurrence and death from any.
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 4.7 | 8.0
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Disease-free survival including ductal carcinoma in situ (DFS-DCIS) in neratinib arm compared to placebo arm; Test type: Other; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.45 to 0.83] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Kaplan-Meier Estimates of Disease-free Survival Including Ductal Carcinoma in Situ (DFS-DCIS) at Year 2 by Treatment Arms
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants | 94.2 [92.6 to 95.4] | 91.3 [89.6 to 92.7]

6. Secondary Outcome: Distant Disease-free Survival (DDFS) in Neratinib Arm Compared to Placebo Arm at Year 2
Description: Distant disease-free survival time is defined as the time from date of randomization until the first occurrence of distant recurrence or death from any cause.
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 3.8 | 5.4
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Distant disease free survival (DDFS) in neratinib arm compared to placebo arm; Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.52 to 1.05] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Kaplan-Meier Estimates of Distant Disease-free Survival (DDFS) at Year 2 by Treatment Arms
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants | 95.3 [93.9 to 96.4] | 94.0 [92.6 to 95.2]

8. Secondary Outcome: Percentage of Participants With Time to Distant Recurrence (TTDR) Event in Neratinib Arm Compared to Placebo Arm at Year 2
Description: Percentage of Participants with TTDR events is reported. TTDR is defined as the time from date of randomization until the first occurrence of distant recurrence or death from breast cancer.
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 3.7 | 5.3
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Time to distant recurrence (TTDR) in neratinib arm compared to placebo arm; Test type: Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.51 to 1.04] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Kaplan-Meier Estimates of Time to Distant Recurrence (TTDR) Survival at Year 2 by Treatment Arms
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants | 95.5 [94.1 to 96.6] | 94.2 [92.8 to 95.3]

10. Secondary Outcome: Central Nervous System Recurrence in Neratinib Arm Compared to Placebo Arm at Year 2
Description: CNS recurrence is defined as the time from randomization to CNS as the first distant recurrence. Competing events include distant recurrence at other sites as the first distant recurrence and death from any cause prior to distant recurrence.
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 0.8 | 1.1

11. Secondary Outcome: Cumulative Incidence of Central Nervous System Recurrence (CNS) at Year 2
Description: Cumulative incidence of Central Nervous System Recurrence (CNS) is estimated by Gray's method (Gray,1988).
Time Frame: From randomization until time of event up to 2 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants | 0.92 [0.49 to 1.59] | 1.16 [0.68 to 1.87]

12. Other Pre Specified Outcome: Invasive Disease-free Survival (iDFS) in Neratinib Arm Compared to Placebo Arm at Year 5
Description: as for outcome 1
Time Frame: From randomization until time of event up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 8.2 | 11.5
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Invasive disease-free survival (iDFS) in neratinib arm compared to placebo arm; Test type: Other; p = 0.008, Log Rank — The Log-rank test is stratified by prior trastuzumab (concurrent or sequential), nodal status (<= 3 or >= 4) and ER/PgR status (positive or negative); Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.92] — [estimate comment as in outcome 1, analysis 1]

13. Other Pre Specified Outcome: Kaplan-Meier Estimates of Invasive Disease-free Survival (iDFS) at Year 5 by Treatment Arms
Time Frame: From randomization until time of event up to 5 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants | 90.2 [88.3 to 91.8] | 87.7 [85.7 to 89.4]

14. Other Pre Specified Outcome: Disease-free Survival Including Ductal Carcinoma in Situ (DFS-DCIS) in Neratinib Arm Compared to Placebo Arm at Year 5
Description: as for outcome 4
Time Frame: From randomization until time of event up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 8.5 | 12.3
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.56 to 0.89] — [estimate comment as in outcome 1, analysis 1]

15. Other Pre Specified Outcome: Distant Disease-free Survival (DDFS) in Neratinib Arm Compared to Placebo Arm at Year 5
Description: as for outcome 6
Time Frame: From randomization until time of event up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 7.0 | 9.2
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.6 to 1.01] — [estimate comment as in outcome 1, analysis 1]

16. Other Pre Specified Outcome: Percentage of Participants With Time to Distant Recurrence (TTDR) Event in Neratinib Arm Compared to Placebo Arm at Year 5
Description: as for outcome 8
Time Frame: From randomization until time of event up to 5 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants with events
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants with events | 6.8 | 8.9
Statistical Analysis 1: Comparison: Neratinib vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.60 to 1.03] — [estimate comment as in outcome 1, analysis 1]

17. Other Pre Specified Outcome: Cumulative Incidence of Central Nervous System Recurrence (CNS) at Year 5
Description: Cumulative incidence of Central Nervous System Recurrence (CNS) is estimated by Gray's method (Gray,1988).
Time Frame: From randomization until time of event up to 5 years
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib | Placebo
Number analyzed (Participants) | 1420 | 1420
percentage of participants | 1.3 [0.77 to 2.06] | 1.82 [1.19 to 2.68]

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after the last dose, up to two years.
Description: The safety population included all participants who received at least one dose of investigational product.
Arm/Group | Neratinib | Placebo
Serious Adverse Events (participants affected / at risk) | 103/1408 | 85/1408
Other Adverse Events (participants affected / at risk) | 1386/1408 | 1234/1408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=1408) | Placebo (N=1408)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 1
Vomiting (Gastrointestinal disorders) | 12 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Rectal cancer (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 3 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Food allergy (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 6 | 4
Erysipelas (Infections and infestations) | 5 | 0
Bronchitis (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 1 | 0
Anorectal cellulitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 4
Rectal abscess (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 3
Diverticulitis (Infections and infestations) | 0 | 1
Incision site cellulitis (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood creatine increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 9 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign female reproductive tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 3 | 2
Ageusia (Nervous system disorders) | 1 | 0
Anosmia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Paresis (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Hyperuricosuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Vulval leukoplakia (Reproductive system and breast disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neratinib (N=1408) | Placebo (N=1408)
Diarrhoea (Gastrointestinal disorders) | 1341 | 499
Nausea (Gastrointestinal disorders) | 605 | 303
Vomiting (Gastrointestinal disorders) | 364 | 113
Abdominal pain (Gastrointestinal disorders) | 339 | 144
Abdominal pain upper (Gastrointestinal disorders) | 212 | 96
Dyspepsia (Gastrointestinal disorders) | 139 | 59
Constipation (Gastrointestinal disorders) | 115 | 134
Stomatitis (Gastrointestinal disorders) | 85 | 29
Abdominal distension (Gastrointestinal disorders) | 73 | 49
Fatigue (General disorders) | 381 | 283
Asthenia (General disorders) | 107 | 110
Pyrexia (General disorders) | 77 | 54
Nasopharyngitis (Infections and infestations) | 84 | 126
Urinary tract infection (Infections and infestations) | 72 | 23
Alanine aminotransferase increased (Investigations) | 118 | 45
Aspartate aminotransferase increased (Investigations) | 101 | 46
Electrocardiogram QT prolonged (Investigations) | 49 | 93
Decreased appetite (Metabolism and nutrition disorders) | 170 | 40
Muscle spasms (Musculoskeletal and connective tissue disorders) | 159 | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 86 | 162
Back pain (Musculoskeletal and connective tissue disorders) | 79 | 134
Pain in extremity (Musculoskeletal and connective tissue disorders) | 58 | 98
Headache (Nervous system disorders) | 278 | 275
Dizziness (Nervous system disorders) | 146 | 127
Insomnia (Psychiatric disorders) | 44 | 73
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 71 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 69 | 92
Rash (Skin and subcutaneous tissue disorders) | 211 | 100
Dry skin (Skin and subcutaneous tissue disorders) | 85 | 33
Hot flush (Vascular disorders) | 40 | 84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less